CLINICAL TRIAL: NCT00580333
Title: A Phase II Trial of Preoperative Cisplatin and Bevacizumab in Estrogen Receptor (ER) Negative, Progesterone (PR) Negative, Human Epidermal Growth Factor Receptor 2 (HER2) Negative Breast Cancer
Brief Title: Preoperative Cisplatin and Bevacizumab in ER-, PR-, HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Steven J Isakoff, MD, PhD, Steven Isakoff, MD, PhD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-202; AVF36335 (Other: Genentech)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: ER negative; PR negative; HER2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin; Bevacizumab; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin/Avastin (Experimental): Cisplatin 75mg/m2 every 3 weeks, neoadjuvant bevacizumab 15mg/m2 every 3 weeks, neoadjuvant doxorubicin, adjuvant (optional) cyclophosphamide , adjuvant (optional) paclitaxel, adjuvant (optional)
  Interventions: Drug: cisplatin; Drug: bevacizumab; Drug: doxorubicin; Drug: cyclophosphamide; Drug: paclitaxel

INTERVENTIONS:
Drug: cisplatin — Preoperatively: Given intravenously on day one of the treatment cycle (once every 3 weeks) for four cycles
  Other Names: platinol
Drug: bevacizumab — Preoperatively: Given intravenously on day 1 of the treatment cycle (once every three weeks) for three cycles Postoperatively: Intravenously for four 2-week cycles (once every two weeks) and after the 8 weeks (study doctor will determine course of treatment) for an additional four 2-week cycles with or with out paclitaxel
  Other Names: Avastin
Drug: doxorubicin — Postoperative: Given intravenously for four 2-week cycles
  Other Names: adriamycin
Drug: cyclophosphamide — Postoperative: Given intravenously for four two-week cycles
  Other Names: cytoxan
Drug: paclitaxel — Postoperative: 8 weeks after postoperative chemotherapy regimen (study doctor will determine course of treatment) paclitaxel for four 2-week cycles (once every two weeks)
  Other Names: taxol

SUMMARY:
The purpose of this study is to find out what effect taking cisplatin in combination with bevacizumab before surgery and then standard chemotherapy plus bevacizumab after surgery will have on participants with Estrogen Receptor (ER) negative, Progesterone Receptor (PR) negative and Human Epidermal Growth Factor Receptor 2 (HER2) negative breast cancer. Cisplatin is used to destroy cancer cells in many types of cancers, and has shown to be effective and have manageable side effects. Bevacizumab is an antibody, which is a protein that attacks a foreign substance in the body. Bevacizumab slows or stops cell growth in cancerous tumors by decreasing the blood supply to the tumors.

DETAILED DESCRIPTION:
* To prepare for surgery, a small "clip" will be placed into the tumor area so that the surgeon can locate the site of the tumor at the time of surgery. This is a standard procedure for breast cancer.
* The study drugs will be given in four 3-week cycles (about 3 months). Participants will come into the clinic each day they receive study treatment intravenously. Cisplatin will be given on day one of the treatment cycle (once every 3 weeks) for four cycles. Bevacizumab will be given on day one of the treatment cycle for three cycles.
* On day one of each 3-week cycle a physical exam, routine blood tests and urine test will be performed. 7-8 days after chemotherapy, blood tests and a hearing test will be performed. A preoperative study visit will take place 7-10 days before surgery and a physical exam, routine blood tests, Electrocardiogram (EKG) and an Magnetic Resonance Imaging (MRI) of the breast will be performed.
* Surgery to remove the tumor will occur at least three weeks after the last dose of cisplatin and is considered standard of care.
* Postoperative chemotherapy will begin at least three weeks after surgery. Everyone on the research study will receive four 2-week cycles of doxorubicin and cyclophosphamide plus bevacizumab. After the 8 weeks, the doctor will decide which of the following two treatment regimens the participant will receive: Bevacizumab for four 2-week cycles (once every two weeks) or; Paclitaxel plus bevacizumab for four 2-week cycles (once every two weeks).
* At the end of the postoperative chemotherapy, the participant will return to the clinic for a medical history, physical exam, vital signs, performance status, routine blood tests, multiple gated acquisition scan (MUGA) or Echocardiogram Scans, and a hearing test.

ELIGIBILITY:
Inclusion Criteria:

* All tumors must be ER-, PR- and HER2-negative
* Clinical stage T2 or T3, N0-3, M0. Subjects with inflammatory breast cancer are not eligible
* For subjects with clinically negative axilla, a sentinel lymph node biopsy will be performed either up front or after preoperative therapy at the discretion of the subject's physicians; for subjects with a clinically positive axilla, a needle aspiration or core biopsy will be performed to confirm the presence of metastatic disease in the lymph nodes.
* 18 years of age or older
* Performance status (PS) of 0 or 1
* Use of an effective means of contraception in subjects of child-bearing potential
* Normal organ function as described in the protocol

Exclusion Criteria:

* Any prior cytotoxic chemotherapy or radiation for the current breast cancer
* HER2-negative ipsilateral breast recurrence, unless prior treatment consisted of excision alone for ductal carcinoma in situ (DCIS)or breast-conserving treatment and hormonal therapy for DCIS or invasive cancer
* Life expectancy of less than 12 weeks
* Current, recent, or planned participation in an experimental durg study other than a Genentech-sponsored bevacizumab cancer study
* Renal dysfunction for which exposure to cisplatin would require dose modifications
* Steroid dependent asthma
* Peripheral neuropathy of any etiology that exceeds grade 1
* Uncontrolled diabetes
* History of malignancy treated without curative intent
* Any other pre-existing medical condition that would represent toxicity in excess of grade 1
* Inadequately controlled hypertension
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive hear failure
* History of myocardial infarction or unstable angina within 12 months prior to study enrollment
* Any history of stroke or transient ischemic attack at any time
* Known central nervous system (CNS) disease
* Significant vascular disease
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 21 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer or bone fracture
* Proteinuria at screening
* Known hypersensitivity to any component of bevacizumab
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula D. Ryan, MD, Principal Investigator — Texas Oncology-The Woodlands
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cisplatin/Avastin
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: stage 2 or 3 triple negative breast cancer
Groups:
- Cisplatin/Avastin: Cisplatin 75mg/m2 every 3 weeks, neoadjuvant bevacizumab 15mg/m2 every 3 weeks, neoadjuvant doxorubicin, adjuvant (optional) cyclophosphamide , adjuvant (optional) paclitaxel, adjuvant (optional)
  cisplatin: Preoperatively: Given intravenously on day one of the treatment cycle (once every 3 weeks) for four cycles
  bevacizumab: Preoperatively: Given IV on day 1 of the treatment cycle (once every three weeks) for three cycles Postoperatively: Intravenously for four 2-week cycles (once every two weeks) and after the 8 weeks (study doctor will determine course of treatment) for an additional four 2-week cycles with or with out paclitaxel
  doxorubicin: Postoperative: Given intravenously for four 2-week cycles
  cyclophosphamide: Postoperative: Given intravenously for four two-week cycles
  paclitaxel: Postoperative: 8 weeks after postoperative chemotherapy regimen (study doctor will determine course of treatment) paclitaxel for four 2-week cycles (once every two weeks)
Arm/Group | Cisplatin/Avastin
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 50 [30 to 66]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate After Preoperative Therapy With Cisplatin and Bevacizumab in ER-, PR-, Human Epidermal Growth Factor Receptor 2 (HER2) -Negative Early Breast Cancer.
Description: The goal of this measure was to determine the pathologic complete response rate (Miller-Payne (MP) score 5) after preoperative therapy with cisplatin and bevacizumab in ER-, PR-, HER2-negative early breast cancer.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cisplatin/Avastin: Cisplatin 75mg/m2 every 3 weeks, neoadjuvant bevacizumab 15mg/m2 every 3 weeks, neoadjuvant doxorubicin, adjuvant (optional) cyclophosphamide , adjuvant (optional) paclitaxel, adjuvant (optional)
  cisplatin: Preoperatively: Given intravenously on day one of the treatment cycle (once every 3 wks) for four cycles
  bevacizumab: Preoperatively: Given intravenously on day 1 of the treatment cycle (once every three wks) for three cycles Postoperatively: Intravenously for four 2-week cycles (once every two weeks) and after the 8 weeks (study doctor will determine course of treatment) for an additional four 2-week cycles with or with out paclitaxel
  doxorubicin: Postoperative: Given intravenously for four 2-week cycles
  cyclophosphamide: Postoperative: Given intravenously for four two-week cycles
  paclitaxel: Postoperative: 8 weeks after postoperative chemotherapy regimen (study doctor will determine course of treatment) paclitaxel for four 2-week cycles (once every two week
Arm/Group | Cisplatin/Avastin
Number analyzed (Participants) | 51
percentage of participants | 16 [7 to 29]

2. Secondary Outcome: Clinical Overall and Complete Response Rates After Preoperative Therapy With Cisplatin and Bevacizumab
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Cisplatin/Avastin: Cisplatin 75mg/m2 every 3 weeks, neoadjuvant bevacizumab 15mg/m2 every 3 weeks, neoadjuvant doxorubicin, adjuvant (optional), cyclophosphamide , adjuvant (optional), paclitaxel, adjuvant (optional)
  cisplatin: Preoperatively: Given intravenously on day one of the treatment cycle (once every 3 weeks) for four cycles
  bevacizumab: Preoperatively: Given intravenously on day 1 of the treatment cycle (once every 3 weeks) for 3 cycles Postoperatively: Intravenously for four 2-week cycles (once every two weeks) and after the 8 weeks (study doctor will determine course of treatment) for an additional four 2-week cycles with or with out paclitaxel
  doxorubicin: Postoperative: Given intravenously for four 2-week cycles
  cyclophosphamide: Postoperative: Given intravenously for four two-week cycles
  paclitaxel: Postoperative: 8 weeks after postoperative chemotherapy regimen (study doctor will determine course of treatment) paclitaxel for four 2-week cycles (once every two week
Arm/Group | Cisplatin/Avastin
Number analyzed (Participants) | 51
Participants
  CR | 12
  OR = CR+PR | 39

3. Secondary Outcome: Toxicity of Administering Bevacizumab in Combination With Standard Adjuvant Chemotherapy.
Description: Number of patients who were unable to receive all cycles of chemotherapy on time for toxicity reasons.
Time Frame: 2 years
Population: analyzed the 43 patients who completed 4 cycles of neoadjuvant therapy and started post-operative treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin/Avastin
Number analyzed (Participants) | 43
Participants | 8

4. Secondary Outcome: Patients With Miller-Payne (MP) Score 3, 4, or 5 Response
Description: To describe a panel of molecular assays for an association with clinical response and, if feasible, with pathologic complete response (pCR) in ER-, PR-, HER2-negative subjects treated with cisplatin and bevacizumab in the preoperative setting. A Miller-Payne (MP) score of 3 indicates a decrease in the size of the cancer by 30% to 90%. A MP score of 4 indicates marked decrease in the size of the cancer by greater than 90%. A MP score of 5 indicates there is no residual cancer remaining (the same as a pathologic complete response).
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cisplatin/Avastin
Number analyzed (Participants) | 51
percentage of participants | 45 [31 to 60]

ADVERSE EVENTS:
Arm/Group | Cisplatin/Avastin
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 51/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin/Avastin (N=51)
fatigue (General disorders) | 36
nausea (Gastrointestinal disorders) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No